CLINICAL TRIAL: NCT01365468
Title: A Phase II Study of RAD001 in the Treatment of Patients With Plexiform Neurofibromas (PN) Associated With Neurofibromatosis Type 1 (NF1)
Brief Title: Efficacy and Safety of RAD001 in Treating Plexiform Neurofibromas (PN) Associated With Neurofibromatosis (NF1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor patients' accrual
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001MIL04T
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Plexiform Neurofibroma Associated With Neurofibromatosis Type 1
Keywords: RAD001,; Everolimus,; Plexiform Neurofibroma,; Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibroma, Plexiform; Neurofibromatosis 1 | interventions — Everolimus

ARMS (1):
- Everolimus (RAD001) (Experimental): enrolled patients received everolimus (RAD001) in an open label manner. Recommended starting dose of everolimus depend on body surface area, starting from 2.5 mg once daily to 7.5 mg once daily.
  Interventions: Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Everolimus (RAD001) — oral daily dosing of tablet starting with 2.5 mg

SUMMARY:
This study was to evaluate the antitumor activity and safety of RAD001 in patients with Plexiform neurofibromas (PN) associated with Neurofibromatosis Type 1 (NF1).

The aim of the study was to :

1. determine whether RAD001, administrated orally daily on a continuous dosing schedule might:

   1. Increases time to disease progression (TTP) based on volumetric MRI measurements in children and adults with NF1 in inoperable documented progressive PN (stratum 1).
   2. Results in objective radiographic responses based on volumetric MRI measurements in children and adults with NF1 and inoperable PN in the absence of documented radiographic progression at the trail entry (stratum
2. To evaluate the tolerability and toxicity of chronic RAD001 administration in this patient population as assessed by the NCI Common Toxicity Criteria, version 4.0.

DETAILED DESCRIPTION:
Approximately 20 patients were to be enrolled to receive everolimus in an open label manner. A total of 9 patients were enrolled to either Stratum 1 or Stratum 2.

The study was open for enrollment up to 2 years. Because the target enrollment was not achieved in this period, study was terminated with less patient than planned.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite diagnosis of NF1 according to the NIH consensus conference criteria.
2. Patients must have PN that have the potential to cause significant morbidity, such as lesions that could compromise the airway or the great vessels, lesions that could cause nerve compression, lesions that could result in major deformity or significant cosmetic problems
3. Measurable disease: patient must have at least one measurable PN amenable to volumetric MRI analysis.

Exclusion Criteria:

1. Chronic treatment with systemic steroids or another immunosuppressive agent.
2. Evidence of an active optic glioma, malignant glioma, malignant peripheral nerve sheath tumor, or other cancer requiring treatment with chemotherapy or radiation therapy.
3. Clinical evidence of significantly impaired lung function
4. Pregnancy or breast feeding.
5. Prior therapy with mTOR inhibitors (e.g.sirolimus, temsirolimus, everolimus).
6. No contraindications for MRI assessments

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Israel (2):
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Litwinsky

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1: Adults and children with neurofibromatosis type 1 (NF1) and inoperable plexiform neurofibromas (PN) with the potential to cause significant morbidity with documented progressive PN prior to study entry wereenrolled in this stratum. Enrolled patients received everolimus (RAD001) in an open label manner. Recommended starting dose of everolimus depend on body surface area, starting from 2.5 mg once daily to 7.5 mg once daily.
- Stratum 2: Adults and children with neurofibromatosis type 1 (NF1) and inoperable plexiform neurofibromas (PN) with the potential to cause significant morbidity that do not have documented progression of the PN at the time of study entry were enrolled in this stratum. Enrolled patients received everolimus (RAD001) in an open label manner. Recommended starting dose of everolimus depend on body surface area, starting from 2.5 mg once daily to 7.5 mg once daily.
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2
Started | 4 | 5
Completed | 0 | 5
Not Completed | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Disease progression | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.7 (14.3) | 16.9 (9.8) | 19.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression (TTP) Based on Change in Volumetric MRI Measurements in Children and Adults (In Stratum I Only)
Description: This endpoint was planned to be analyzed for only Stratum 1 patients. Progression of disease defined as a ≥ 20% increase in the volume (by volumetric MRI) of at least one of the index plexiform neurofibromas (PN) compared to the pretreatment volume measured prior to the start of the current treatment phase.
Time Frame: Screening, after course #6, #12, #18, #24, End of Treatment(1 course=28days)
Population: The Full Analysis Set (FAS) consisted of all enrolled patients.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Stratum 1
Number analyzed (Participants) | 4
Days | NA [NA to NA] — Median was not achieved because only one progression event occurred.

2. Primary Outcome: Number of Patients With Objective Radiographic Responses Based on Volumetric MRI Measurements (In Stratum 2 Only)
Description: Response was assessed at the time that a follow up volumetric MRI scan is performed (after course 6 and then every 6 months and at the end of treatment).
  * Complete response (CR): complete resolution of all measurable or palpable PN for ≥ 28days and no appearance of new lesions.
  * Partial response (PR): A ≥ 20% reduction in the sum of the volume of all index PN lesions for ≥ 28days.
  * Stable disease (SD): A < 20% increase and < 20% decrease in the sum of the volume of all index PN lesions for ≥ 28days.
Time Frame: Screening, after course #6, then every 6 months and end of treatment(1 course=28days)
Population: The Full Analysis Set (FAS) consisted of all enrolled patients.
Measure: Number; unit: Patients
Arm/Group | Stratum 2
Number analyzed (Participants) | 5
Patients
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 5

3. Primary Outcome: Number of Patients With Adverse Events Assessed by Common Toxicity Criteria for Adverse Events (CTCAE) V.04
Description: Adverse events were assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0. If CTCAE grading does not exist for an adverse event, the severity of mild, moderate, severe, and life-threatening, corresponding to grades 1 - 4 respectively, were used. CTCAE grade 5 (death) was not used in this study.
Time Frame: From the time ICF was signed until 28 days after End of Treatment (up to a maximum of 25 months)
Population: The Safety Population consisted of all patients who received at least one dose of study treatment and had at least one post-baseline safety assessment.
Measure: Number; unit: Patients
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 4 | 5
Patients
  At least one Grade 1 AE | 4 | 5
  At least one Grade 2 AE | 4 | 5
  At least one Grade 3 AE | 1 | 0
  At least one Grade 4 AE | 1 | 0

4. Other Pre Specified Outcome: Number of Patients With Clinical Response
Description: Clinical response is defined as improvement of function, performance status, or decrease in PN related pain persisting for at least 28 days on treatment.
Time Frame: Screening, Day 1, after course #3, #6, #12, #18, #24, End of Treatment (1 course = 28 days)
Population: Study got terminated because of poor patient's accrual. Enrolled patients were less than planned number of patients required for analysis. Hence, planned analysis was not done.
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Physician's Global Assessment of Clinical Condition (PGA) of Skin Lesions
Description: The Physician"s Global Assessment of Clinical Condition (PGA) is a 7-point grading scale for the investigator's assessment of the overall extent of improvement or worsening of the patient"s skin disease as compared to baseline. Responses must be confirmed by at least two assessments separated in time by at least 4 weeks. The grading ranges from 0 to 6; 0 is Completely clear where as 6 is for worse condition. A complete clinical response (CCR) requires a grading of 0 indicating the absence of disease (histological confirmation is not required). Grades 1, 2, and 3 constitute partial response, indicating improvement of at least 50 percent, but less than 100 percent improvement.
Time Frame: Screening, after course #3, #6, #12, #18, #24, End of Treatment (1 course = 28 days)
Population: as for outcome 4
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Stratum 1 | Stratum 2
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 (N=4) | Stratum 2 (N=5)
Hypersensitivity (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 (N=4) | Stratum 2 (N=5)
Ear pain (Ear and labyrinth disorders) | 2 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
Influenza like illness (General disorders) | 3 | 1
Mucosal inflammation (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tendonitis (Injury, poisoning and procedural complications) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 1
Drug level increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 4
Paraesthesia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Tic (Psychiatric disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Cytoreductive surgery (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
Study got terminated because of poor patient's accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.